CLINICAL TRIAL: NCT03387137
Title: Phase I Placebo-Controlled Study of the Infectivity, Safety and Immunogenicity of a Single Dose of a Recombinant Live-Attenuated Respiratory Syncytial Virus Vaccine, RSV 6120/∆NS2/1030s, Lot RSV#012A, Delivered as Nose Drops to RSV-Seropositive Children 12 to 59 Months of Age and RSV-Seronegative Infants and Children 6 to 24 Months of Age
Brief Title: Evaluating the Infectivity, Safety, and Immunogenicity of a Respiratory Syncytial Virus Vaccine (RSV 6120/∆NS2/1030s) in RSV-Seropositive Children and RSV-Seronegative Infants and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 322
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: RSV 6120/∆NS2/1030s Vaccine (Experimental): RSV-seropositive children will receive a single dose of 10^5.7 plaque-forming units (PFUs) of RSV 6120/∆NS2/1030s vaccine at study entry (Day 0).
  Interventions: Biological: RSV 6120/∆NS2/1030s
- Group 1: Placebo (Placebo Comparator): RSV-seropositive children will receive a single dose of placebo at study entry (Day 0).
  Interventions: Biological: Placebo
- Group 2: RSV 6120/∆NS2/1030s Vaccine (Experimental): RSV-seronegative infants and children will receive a single dose of 10^5.0 PFUs of RSV 6120/∆NS2/1030s vaccine at study entry (Day 0).
  Interventions: Biological: RSV 6120/∆NS2/1030s
- Group 2: Placebo (Placebo Comparator): RSV-seronegative infants and children will receive a single dose of placebo at study entry (Day 0).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSV 6120/∆NS2/1030s — Delivered as nose drops
  Arms: Group 1: RSV 6120/∆NS2/1030s Vaccine; Group 2: RSV 6120/∆NS2/1030s Vaccine
Biological: Placebo — Delivered as nose drops
  Arms: Group 1: Placebo; Group 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the infectivity, safety, and immunogenicity of a single dose of a recombinant, live-attenuated respiratory syncytial virus (RSV) vaccine (RSV 6120/∆NS2/1030s) in RSV-seropositive children 12 to 59 months of age and RSV-seronegative infants and children 6 to 24 months of age.

DETAILED DESCRIPTION:
This study will evaluate the infectivity, safety, and immunogenicity of a single dose of a recombinant, live-attenuated RSV vaccine (RSV 6120/∆NS2/1030s) in RSV-seropositive children 12 to 59 months of age and RSV-seronegative infants and children 6 to 24 months of age.

The vaccine will be evaluated in a stepwise fashion beginning in RSV-seropositive children (Group 1), and then in RSV-seronegative infants and children (Group 2). In each group, participants will be randomly assigned to receive a single dose of RSV 6120/∆NS2/1030s vaccine or placebo at study entry (Day 0).

Participants will be enrolled in the study between April 1 and October 31, outside of the RSV season. Group 1 (RSV-seropositive children) will be followed for 28 days. Group 2 (RSV-seronegative infants and children) will remain on study until they complete the post-RSV season visit.

Group 2 participants may participate in an optional second season of RSV surveillance during November to March of the second year following enrollment.

Study visits for all participants may include clinical assessments, blood collection, and nasal washes. Additionally, participants' parents or guardians will be contacted by study staff at various times during the study to monitor participants' health.

ELIGIBILITY:
Inclusion Criteria for RSV-Seropositive Children:

* Greater than or equal to 12 months of age and less than 60 months of age at the time of inoculation
* Screening serum specimen for RSV neutralizing antibody is obtained within the calendar year of inoculation
* Seropositive for RSV antibody, defined as serum RSV neutralizing antibody titer greater than or equal to 1:40
* Pre-inoculation serum sample for RSV neutralizing antibody testing is obtained no more than 56 days prior to inoculation
* In good health based on review of the medical record, history, and physical examination at the time of inoculation
* Received routine immunizations appropriate for age based on the Advisory Committee on Immunization Practices (ACIP) Recommended Immunization Schedule for Children and Adolescents Aged 18 Years or Younger
* Growing normally for age as demonstrated on a standard growth chart and has a current height and weight above the 3rd percentile for age
* Expected to be available for the duration of the study
* Parent/guardian is willing and able to provide written informed consent

Exclusion Criteria for RSV-Seropositive Children:

* Born at less than 34 weeks gestation
* Maternal history of positive HIV test
* Evidence of chronic disease
* Known or suspected impairment of immune function
* Bone marrow/solid organ transplant recipient
* Major congenital malformations, including congenital cleft palate or cytogenetic abnormalities
* Suspected or documented developmental disorder, delay, or other developmental problem
* Cardiac abnormality requiring treatment
* Lung disease or reactive airway disease
* More than one episode of wheezing in the first year of life
* Wheezing episode or received bronchodilator therapy within the past 12 months
* Wheezing episode or received bronchodilator therapy after the age of 12 months
* Previous receipt of supplemental oxygen therapy in a home setting
* Previous receipt of an investigational RSV vaccine
* Previous receipt or planned administration of anti-RSV drug (ribavirin) or RSV antibody product including RSV immune globulin (RSV Ig) or RSV monoclonal antibody (RSV mAb)
* Previous receipt of immunoglobulin or any antibody products within the past 6 months
* Previous receipt of any other blood products within the past 6 months
* Previous anaphylactic reaction
* Previous vaccine-associated adverse reaction that was Grade 3 or above
* Known hypersensitivity to any vaccine component
* Member of a household that contains an infant who is less than 12 months of age at the date of inoculation through the 10th day after inoculation
* Member of a household that, at the date of inoculation through the 10th day after inoculation, contains an immunocompromised individual including but not limited to:

  * a person who is HIV-infected
  * a person who has received chemotherapy within the 12 months prior to enrollment
  * a person receiving immunosuppressant agents
  * a person living with a solid organ or bone marrow transplant
* Will attend a daycare facility that does not separate children by age and contains an infant who is less than 12 months of age at the date of inoculation through the 10th day after inoculation
* Receipt of any of the following prior to enrollment:

  * any inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days prior, or
  * any live vaccine, other than rotavirus vaccine, within the 28 days prior, or
  * another investigational vaccine or investigational drug within 28 days prior, or
  * salicylate (aspirin) or salicylate-containing products within the past 28 days
* Scheduled administration of any of the following after planned inoculation:

  * inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days after, or
  * any live vaccine other than rotavirus in the 28 days after, or
  * another investigational vaccine or investigational drug in the 28 days after
* Receipt of any of the following medications within 3 days of study enrollment:

  * systemic antibacterial, antiviral, antifungal, anti-parasitic, or antituberculous agents, whether for treatment or prophylaxis, or
  * intranasal medications, or
  * other prescription medications except the permitted concomitant medications listed below:
  * Permitted concomitant medications (prescription or non-prescription) include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including (but not limited to) cutaneous (topical) steroids, topical antibiotics, and topical antifungal agents.
* Any of the following events at the time of enrollment:

  * fever (temporal or rectal temperature of greater than or equal to 100.4°F), or
  * upper respiratory signs or symptoms (rhinorrhea, cough, or pharyngitis) or
  * nasal congestion significant enough to interfere with successful inoculation, or
  * otitis media

Inclusion Criteria for RSV-Seronegative Infants and Children:

* Greater than or equal to 6 months of age and less than 25 months of age at the time of inoculation
* Screening and pre-inoculation serum specimens for RSV-neutralizing antibody are obtained no more than 42 days prior to inoculation
* Seronegative for RSV antibody, defined as serum RSV-neutralizing antibody titer less than 1:40
* In good health based on review of the medical record, history, and physical examination at the time of inoculation
* Received routine immunizations appropriate for age based on the ACIP Recommended Immunization Schedule for Children and Adolescents Aged 18 Years or Younger
* Growing normally for age as demonstrated on a standard growth chart, AND

  * If less than 1 year of age: has a current height and weight above the 5th percentile for age
  * If greater than or equal to 1 year of age: has a current height and weight above the 3rd percentile for age
* Expected to be available for the duration of the study
* Parent/guardian is willing and able to provide written informed consent

Exclusion Criteria for RSV-Seronegative Infants and Children:

* Born at less than 34 weeks gestation
* Born at less than 37 weeks gestation, and at the date of inoculation less than 1 year of age
* Maternal history of a positive HIV test
* Evidence of chronic disease
* Known or suspected infection or impairment of immunological functions
* Bone marrow/solid organ transplant recipient
* Major congenital malformations, including congenital cleft palate or cytogenetic abnormalities
* Suspected or documented developmental disorder, delay, or other developmental problem
* Cardiac abnormality requiring treatment
* Lung disease or reactive airway disease
* More than one episode of wheezing in the first year of life
* Wheezing episode or received bronchodilator therapy within the past 12 months
* Wheezing episode or received bronchodilator therapy after the age of 12 months
* Previous receipt of supplemental oxygen therapy in a home setting
* Previous receipt of an investigational RSV vaccine
* Previous receipt or planned administration of anti-RSV antibody product including ribavirin, RSV Ig, or RSV mAb
* Previous receipt of immunoglobulin or any antibody products within the past 6 months
* Previous receipt of any blood products within the past 6 months
* Previous anaphylactic reaction
* Previous vaccine-associated adverse reaction that was Grade 3 or above
* Known hypersensitivity to any study product component
* Member of a household that contains an infant who is less than 6 months of age at the date of inoculation through the 28th day after inoculation
* Member of a household that, at the date of inoculation through the 28th day after inoculation, contains an immunocompromised individual including but not limited to:

  * a person who is HIV-infected
  * a person who has cancer and has received chemotherapy within the 12 months prior to enrollment
  * a person living with a solid organ or bone marrow transplant
* Attends a daycare facility that does not separate children by age and contains an infant less than 6 months of age at the date of inoculation through the 28th day after inoculation
* Receipt of any of the following prior to enrollment:

  * any inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days prior, or
  * any live vaccine, other than rotavirus vaccine, within the 28 days prior, or
  * another investigational vaccine or investigational drug within 28 days prior, or
  * salicylate (aspirin) or salicylate-containing products within the past 28 days
* Scheduled administration of any of the following after planned inoculation

  * inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days after, or
  * any live vaccine other than rotavirus in the 28 days after, or
  * another investigational vaccine or investigational drug in the 56 days after
* Receipt of any of the following medications within 3 days of study enrollment:

  * systemic antibacterial, antiviral, antifungal, anti-parasitic, or antituberculous agents, whether for treatment or prophylaxis, or
  * intranasal medications, or
  * other prescription medications except the permitted concomitant medications listed below:
  * Permitted concomitant medications (prescription or non-prescription) include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including (but not limited to) cutaneous (topical) steroids, topical antibiotics, and topical antifungal agents.
* Any of the following events at the time of enrollment:

  * fever (temporal or rectal temperature of greater than or equal to 100.4°F), or
  * upper respiratory signs or symptoms (rhinorrhea, cough, or pharyngitis) or
  * nasal congestion significant enough to interfere with successful inoculation, or
  * otitis media

Inclusion Criteria for RSV-Seronegative Children Participating in a Second Season of RSV Surveillance:

* RSV-seronegative participants who have completed the initial RSV season surveillance portion of the study and whose parent/guardian is willing and able to provide written informed consent
* Expected to be available during the second year of RSV surveillance

Exclusion Criteria for RSV-Seronegative Children Participating in a Second Season of RSV Surveillance:

* Currently enrolled in another RSV study

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health (JHSPH)
Locations (1):
- Center for Immunization Research, Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Result] Karron RA, Luongo C, Woods S, Oliva J, Collins PL, Buchholz UJ; RSVPed Team. Evaluation of the Live-Attenuated Intranasal Respiratory Syncytial Virus (RSV) Vaccine RSV/6120/DeltaNS2/1030s in RSV-Seronegative Young Children. J Infect Dis. 2024 Feb 14;229(2):346-354. doi: 10.1093/infdis/jiad281. PMID 37493269

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from pediatric practices and clinics in the greater Baltimore/Washington area based on referral by the primary care provider or the provider's staff; and through mailing IRB-approved documents to children of local pediatric practices and clinics, and to households in local zip codes containing age-appropriate children between September 2017 and September 2019. The first participant was enrolled on 10/13/2017 and the last participant was enrolled on 9/27/2019.
Pre-assignment Details: Of the 73 participants that were screened, 45 met eligibility criteria, parent agreed to enroll and were inoculated with study product.
Period: Overall Study
Arm/Group | Group 1: RSV 6120/∆NS2/1030s Vaccine | Group 1: Placebo | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Started | 10 | 5 | 20 | 10
Completed | 10 | 5 | 20 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: RSV 6120/∆NS2/1030s Vaccine | Group 1: Placebo | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo | Total
Number analyzed (Participants) | 10 | 5 | 20 | 10 | 45
Age, Customized [Count of Participants; unit: Participants] — Group 1 enrolled children 12-59 months of age. Group 2 enrolled infants and children 6-24 months of age.
  Participants
    < 1 year of age | 0 | 0 | 7 | 5 | 12
    1 year of age | 6 | 1 | 12 | 5 | 24
    2 years of age | 1 | 2 | 1 | 0 | 4
    3 years of age | 2 | 0 | 0 | 0 | 2
    4 years of age | 1 | 2 | 0 | 0 | 3
    > 4 years of age | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 11 | 3 | 24
  Male | 4 | 1 | 9 | 7 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 10 | 5 | 18 | 10 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 6 | 1 | 16 | 9 | 32
  More than one race | 1 | 3 | 2 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 20 | 10 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Events (AEs) by Grade - (RSV-seropositive Participants)
Description: Solicited adverse events include fever; otitis media; upper respiratory illness (URI); lower respiratory illness (LRI) and cough (without LRI) as defined in Appendix IV of the protocol document. The number of participants who experienced solicited adverse events was presented. A participant was only counted once in each solicited AE category, and that is in the line corresponding to the highest grade adverse event they had in that category. These events were graded (Grade 1-mild to Grade 4-life-threatening) following protocol-defined grading system outlined in Table 21 and Table 22 in the protocol document.
Time Frame: Measured through Day 10
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: RSV 6120/∆NS2/1030s Vaccine | Group 1: Placebo
Number analyzed (Participants) | 10 | 5
Participants
  Fever: Did not have this AE | 8 | 5
  Fever: Grade 1 | 0 | 0
  Fever: Grade 2 | 2 | 0
  Fever: Grade 3 | 0 | 0
  Fever: Grade 4 | 0 | 0
  Upper Respiratory Illness (URI): Did not have this AE | 6 | 4
  Upper Respiratory Illness (URI): Grade 1 | 4 | 1
  Upper Respiratory Illness (URI): Grade 2 | 0 | 0
  Upper Respiratory Illness (URI): Grade 3 | 0 | 0
  Upper Respiratory Illness (URI): Grade 4 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Did not have this AE | 10 | 5
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 1 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 2 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 3 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 4 | 0 | 0
  LRI in the absence of RSV shedding: Did not have this AE | 9 | 5
  LRI in the absence of RSV shedding: Grade 1 | 0 | 0
  LRI in the absence of RSV shedding: Grade 2 | 1 | 0
  LRI in the absence of RSV shedding: Grade 3 | 0 | 0
  LRI in the absence of RSV shedding: Grade 4 | 0 | 0
  Cough without LRI: Did not have this AE | 9 | 5
  Cough without LRI: Grade 1 | 1 | 0
  Cough without LRI: Grade 2 | 0 | 0
  Cough without LRI: Grade 3 | 0 | 0
  Cough without LRI: Grade 4 | 0 | 0
  Otitis Media: Did not have this AE | 10 | 5
  Otitis Media: Grade 1 | 0 | 0
  Otitis Media: Grade 2 | 0 | 0
  Otitis Media: Grade 3 | 0 | 0
  Otitis Media: Grade 4 | 0 | 0

2. Primary Outcome: Number of Participants With Solicited Adverse Events (AEs) by Grade - (RSV-seronegative Participants)
Description: Solicited adverse events include fever; otitis media; upper respiratory illness (URI); lower respiratory illness (LRI) and cough (without LRI) as defined by Appendix IV in the protocol document . The number of participants who experienced solicited adverse events was presented. A participant was only counted once in each solicited AE category, and that is in the line corresponding to the highest grade adverse event they had in that category. These events were graded (Grade 1-mild to Grade 4-life-threatening) following protocol-defined grading system outlined in Table 21 and Table 22 in the protocol document.
Time Frame: Measured through Day 28
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Number analyzed (Participants) | 20 | 10
Participants
  Fever: Did not have this AE | 14 | 8
  Fever: Grade 1 | 1 | 1
  Fever: Grade 2 | 4 | 1
  Fever: Grade 3 | 1 | 0
  Fever: Grade 4 | 0 | 0
  Upper Respiratory Illness (URI): Did not have this AE | 2 | 6
  Upper Respiratory Illness (URI): Grade 1 | 18 | 4
  Upper Respiratory Illness (URI): Grade 2 | 0 | 0
  Upper Respiratory Illness (URI): Grade 3 | 0 | 0
  Upper Respiratory Illness (URI): Grade 4 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Did not have this AE | 19 | 10
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 1 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 2 | 1 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 3 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 4 | 0 | 0
  LRI in the absence of RSV shedding: Did not have this AE | 19 | 10
  LRI in the absence of RSV shedding: Grade 1 | 0 | 0
  LRI in the absence of RSV shedding: Grade 2 | 1 | 0
  LRI in the absence of RSV shedding: Grade 3 | 0 | 0
  LRI in the absence of RSV shedding: Grade 4 | 0 | 0
  Cough, without LRI: Did not have this AE | 14 | 9
  Cough, without LRI: Grade 1 | 5 | 1
  Cough, without LRI: Grade 2 | 1 | 0
  Cough, without LRI: Grade 3 | 0 | 0
  Cough, without LRI: Grade 4 | 0 | 0
  Otitis Media: Did not have this AE | 19 | 10
  Otitis Media: Grade 1 | 0 | 0
  Otitis Media: Grade 2 | 1 | 0
  Otitis Media: Grade 3 | 0 | 0
  Otitis Media: Grade 4 | 0 | 0

3. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs) - (RSV-seropositive Participants)
Description: Unsolicited adverse events were other events, not included in the solicited AEs. The number of participants who experienced unsolicited adverse events was presented.
Time Frame: Measured through Day 10
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: RSV 6120/∆NS2/1030s Vaccine | Group 1: Placebo
Number analyzed (Participants) | 10 | 5
Participants | 3 | 1

4. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs) - (RSV-seronegative Participants)
Description: as for outcome 3
Time Frame: Measured through Day 28
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Number analyzed (Participants) | 20 | 10
Participants | 9 | 3

5. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) (RSV-seropositive Participants)
Description: A Serious Adverse Event (SAE) is an AE, whether considered related to the study product or not, that:
  * Results in death during the period of protocol-defined surveillance;
  * Is life threatening: defined as an event in which the patient was at immediate risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death were it more severe;
  * Requires inpatient hospitalization (or prolongation of existing hospitalization): defined as at least an overnight stay in the hospital or emergency ward for treatment that would have been inappropriate if administered in the outpatient setting;
  * Results in a persistent or significant disability/incapacity;
  * Is a congenital anomaly or birth defect, OR
  * Is an important medical event that may not be immediately life threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the outcomes listed above.
Time Frame: Measured through Day 28
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: RSV 6120/∆NS2/1030s Vaccine | Group 1: Placebo
Number analyzed (Participants) | 10 | 5
Participants | 0 | 0

6. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) (RSV-seronegative Participants)
Description: as for outcome 5
Time Frame: Measured through Day 56
Population: Study participants who received inoculation and were followed on study pst Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Number analyzed (Participants) | 20 | 10
Participants | 0 | 0

7. Primary Outcome: Frequency of Infection With RSV Vaccine Virus (RSV-seropositive Subjects)
Description: As defined as 1) vaccine virus identified in a nasal wash (a binary outcome based on nasal washes done throughout the study period; Day 0 nasal wash will be counted as baseline) and/or 2) a greater than or equal to 4-fold rise in RSV neutralizing antibody titer and/or serum enzyme-linked immunosorbent assay (ELISA) titer to the RSV F protein from study entry to Study Day 28.
Time Frame: Measured through Day 28
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: RSV 6120/∆NS2/1030s Vaccine | Group 1: Placebo
Number analyzed (Participants) | 10 | 5
Participants | 2 | 0

8. Primary Outcome: Frequency of Infection With RSV Vaccine Virus (RSV-seronegative Subjects)
Description: As defined as 1) vaccine virus identified in a nasal wash (a binary outcome based on nasal washes done throughout the study period; Day 0 nasal wash will be counted as baseline) and/or 2) a greater than or equal to 4-fold rise in RSV neutralizing antibody titer and/or serum enzyme-linked immunosorbent assay (ELISA) titer to the RSV F protein from study entry to Study Day 56.
Time Frame: Measured through Day 56
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Number analyzed (Participants) | 20 | 10
Participants | 20 | 0

9. Primary Outcome: Peak Titer of Vaccine Virus Shed Measured by Culture (RSV-seropositive Subjects)
Description: This is the mean of the highest value per participant of the titer of vaccine virus shed. It was measured by culture. Only participants who met the definition of infection with vaccine virus were included.
Time Frame: Measured at Days 0, 3, 4, 5, 6, 7 and 10
Population: Only participants who met the definition of infection with vaccine virus were included.
Measure: Mean (Standard Deviation); unit: log 10 PFU/mL
Arm/Group | Group 1: RSV 6120/∆NS2/1030s Vaccine | Group 1: Placebo
Number analyzed (Participants) | 2 | 0
log 10 PFU/mL | 1.2 (0.5) |

10. Primary Outcome: Peak Titer of Vaccine Virus Shed Measured by Reverse Transcription Polymerase Chain Reaction (RSV-seropositive Subjects)
Description: This is the mean of the highest value per participant of the titer of vaccine virus shed. It was measured by reverse transcription polymerase chain reaction (RT-PCR). Only participants who met the definition of infection with vaccine virus were included.
Time Frame: Measured at Days 0, 3, 4, 5, 6, 7 and 10
Population: Only participants who met the definition of infection with vaccine virus were included.
Measure: Mean (Standard Deviation); unit: log 10 copies/mL
Arm/Group | Group 1: RSV 6120/∆NS2/1030s Vaccine | Group 1: Placebo
Number analyzed (Participants) | 2 | 0
log 10 copies/mL | 3.1 (0.9) |

11. Primary Outcome: Duration of Vaccine Virus Shedding in Nasal Washes (RSV-seropositive Subjects)
Description: As determined by a) culture and b) reverse transcription polymerase chain reaction (RT-PCR)
Time Frame: Measured at Days 0, 3, 4, 5, 6, 7 and 10. Last day positive is reported.
Population: Only participants who met the definition of infection with vaccine virus were included.
Measure: Mean (Full Range); unit: Days
Arm/Group | Group 1: RSV 6120/∆NS2/1030s Vaccine | Group 1: Placebo
Number analyzed (Participants) | 2 | 0
Days
  Culture Positive | 7.5 [5 to 10] |
  RT-PCR Positive | 7.5 [5 to 10] |

12. Primary Outcome: Peak Titer of Vaccine Virus Shed by Culture (RSV-seronegative Subjects)
Description: as for outcome 9
Time Frame: Measured at Days 0, 3, 5, 7, 10, 12, 14, 17 and 28
Population: Only participants who met the definition of infection with vaccine virus were included.
Measure: Mean (Standard Deviation); unit: log 10 PFU/mL
Arm/Group | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Number analyzed (Participants) | 20 | 0
log 10 PFU/mL | 3.0 (0.8) |

13. Primary Outcome: Peak Titer of Vaccine Virus Shed by Reverse Transcription Polymerase Chain Reaction (RSV-seronegative Subjects)
Description: as for outcome 10
Time Frame: Measured at Days 0, 3, 5, 7, 10, 12, 14, 17 and 28
Population: Only participants who met the definition of infection with vaccine virus were included.
Measure: Mean (Standard Deviation); unit: log 10 copies/mL
Arm/Group | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Number analyzed (Participants) | 20 | 0
log 10 copies/mL | 4.5 (0.8) |

14. Primary Outcome: Duration of Vaccine Virus Shedding in Nasal Washes (RSV-seronegative Subjects)
Description: As determined by a) culture and b) reverse transcription polymerase chain reaction (RT-PCR)
Time Frame: Measured at Days 0, 3, 5, 7, 10, 12, 14, 17 and 28. Lat day positive is reported
Population: Only participants who met the definition of infection with vaccine virus were included.
Measure: Mean (Full Range); unit: Days
Arm/Group | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Number analyzed (Participants) | 20 | 0
Days
  Culture Positive | 10.2 [7 to 14] |
  RT-PCR Positive | 11.8 [7 to 17] |

15. Primary Outcome: Number of Participants With a Greater Than or Equal to 4-fold Rise in Serum RSV-neutralizing Antibody Titers and/or Serum Antibody Titers to RSV F Glycoprotein(RSV-seropositive Subjects)
Description: Serum RSV-neutralizing antibody titers were assessed by 60% RSV-plaque reduction neutralization titer (RSV-PRNT) assay and an Enzyme-linked Immunosorbent Assay (ELISA). Antibody responses were defined as a greater than or equal to 4-fold increase in titer in paired specimens, between pre-inoculation and post-inoculation time points.
Time Frame: Measured at Day 0 and Day 28
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: RSV 6120/∆NS2/1030s Vaccine | Group 1: Placebo
Number analyzed (Participants) | 10 | 5
Participants
  Serum RSV Neutralizing Antibody Titers | 0 | 0
  Serum IgG ELISA RSV F Antibody Interpolated Titers | 0 | 0

16. Primary Outcome: Number of Participants With a Greater Than or Equal to 4-fold Rise in Serum RSV-neutralizing Antibody Titers and/or Serum Antibody Titers to RSV F Glycoprotein (RSV-seronegative Subjects)
Description: as for outcome 15
Time Frame: Measured at Day 0 and Day 56
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Number analyzed (Participants) | 20 | 10
Participants
  Serum RSV Neutralizing Antibody Titers | 18 | 0
  Serum IgG ELISA RSV F Antibody Interpolated Titers | 17 | 0

17. Primary Outcome: RSV-neutralizing Serum Antibody Titer and Immunoglobulin G (IgG) Serum Antibody Titers to RSV F Glycoprotein Enzyme-linked Immunosorbent Assay (ELISA)(RSV-seropositive Subjects)
Description: Serum RSV-neutralizing antibody titers were assessed by 60% RSV-plaque reduction neutralization titer (RSV-PRNT) assay. Serum antibody titers to RSV F glycoprotein were assessed by ELISA.
Time Frame: Measured at Day 28
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Mean (Standard Deviation); unit: log 2 titers
Arm/Group | Group 1: RSV 6120/∆NS2/1030s Vaccine | Group 1: Placebo
Number analyzed (Participants) | 10 | 5
log 2 titers
  Serum RSV Neutralizing Antibody Titers | 7.1 (1.0) | 7.2 (0.7)
  Serum IgG ELISA RSV F Antibody Interpolated Titers | 12.1 (1.5) | 12.9 (0.5)

18. Primary Outcome: RSV-neutralizing Serum Antibody Titers and Immunoglobulin G (IgG) Serum Antibody Titers to RSV F Glycoprotein Enzyme-linked Immunosorbent Assay (ELISA) (RSV-seronegative Subjects)
Description: as for outcome 17
Time Frame: Measured at Day 56
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Mean (Standard Deviation); unit: log 2 titers
Arm/Group | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Number analyzed (Participants) | 20 | 10
log 2 titers
  Serum RSV Neutralizing Antibody Titers | 6.5 (1.1) | 2.6 (0.6)
  Serum IgG ELISA RSV F Antibody Interpolated Titers | 10.9 (1.7) | 6.0 (2.0)

19. Secondary Outcome: Number of RSV-seronegative (Group 2) Vaccine and Placebo Recipients Who Experience Natural Infection With wt RSV During the First RSV Season
Description: As defined as 1) RSV identified in a nasal wash (a binary outcome based on nasal washes done throughout the RSV surveillance period; or 2) a greater than or equal to 4-fold rise in RSV neutralizing antibody titer or Serum IgG RSV F antibody titer from pre- to post-RSV Surveillance season
Time Frame: Measured through participants' last study visit, up to a total of 6 to 13 months after study entry, depending on when participants enrolled in the study.
Population: Only participants who had RSV detected in nasal washes or had greater than or equal to 4 fold rise in serum antibodies from pre- to post-RSV season in the absence of RSV-associated medical events were included.
  Four vaccinees and 2 placebo recipients were excluded due to SARS CoV-2 pandemic and no post-surveillance sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Number analyzed (Participants) | 16 | 8
Participants | 6 | 5

20. Secondary Outcome: Frequency of Symptomatic, Medically Attended Respiratory and Febrile Illness in the RSV-seronegative (Group 2) Vaccine and Placebo Recipients Who Experience Natural Infection With wt RSV During the First RSV Season
Description: The number of participants who had RSV-associated, symptomatic, medically attended respiratory and febrile illness (MAARI) among those who had indicators of natural infection with wt RSV were presented. Natural infection with wt RSV during the RSV season surveillance was defined as having either RSV detected in nasal washes collected during illness visits for MAARI events or a > 4-fold rise in serum antibodies from pre- to post-RSV season in the absence of RSV-associated medical events.
Time Frame: Measured through participants' last study visit, up to a total of 6 to 13 months after study entry, depending on when participants enroll in the study.
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Number analyzed (Participants) | 6 | 5
Participants | 4 | 3

21. Secondary Outcome: Severity of Symptomatic, Medically Attended Respiratory and Febrile Illness in the RSV-seronegative (Group 2) Vaccine and Placebo Recipients Who Experience Natural Infection With wt RSV During the First RSV Season
Description: The number of participants who had RSV-associated, symptomatic, medically attended respiratory and febrile illness (MAARI) among those who had indicators of natural infection with wt RSV were presented. Natural infection with wt RSV during the RSV season surveillance was defined as having either RSV detected in nasal washes collected during illness visits for MAARI events or a > 4-fold rise in serum antibodies from pre- to post-RSV season in the absence of RSV-associated medical events. A participant was only counted once in each MAARI category, and that was in the line corresponding to the highest grade adverse event they had in that category. These events were graded (Grade 1-mild to Grade 4-life-threatening) following protocol-defined grading system outlined in Table 21 and Table 22 in the protocol document.Assessed by protocol-determined grading system
Time Frame: as for outcome 20
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Number analyzed (Participants) | 6 | 5
Participants
  Medically Attended Fever: No adverse event | 3 | 3
  Medically Attended Fever: Grade 1 | 0 | 0
  Medically Attended Fever: Grade 2 | 1 | 1
  Medically Attended Fever: Grade 3 | 2 | 1
  Medically Attended Fever: Grade 4 | 0 | 0
  Medically Attended URI: No adverse event | 2 | 1
  Medically Attended URI: Grade 1 | 0 | 0
  Medically Attended URI: Grade 2 | 4 | 4
  Medically Attended URI: Grade 3 | 0 | 0
  Medically Attended URI: Grade 4 | 0 | 0
  Medically Attended LRI: No adverse event | 4 | 5
  Medically Attended LRI: Grade 1 | 0 | 0
  Medically Attended LRI: Grade 2 | 2 | 0
  Medically Attended LRI: Grade 3 | 0 | 0
  Medically Attended LRI: Grade 4 | 0 | 0
  Medically Attended Cough: No adverse event | 3 | 2
  Medically Attended Cough: Grade 1 | 0 | 0
  Medically Attended Cough: Grade 2 | 3 | 3
  Medically Attended Cough: Grade 3 | 0 | 0
  Medically Attended Cough: Grade 4 | 0 | 0
  Medically Attended Otitis Media: No adverse event | 4 | 4
  Medically Attended Otitis Media: Grade 1 | 0 | 0
  Medically Attended Otitis Media: Grade 2 | 2 | 1
  Medically Attended Otitis Media: Grade 3 | 0 | 0
  Medically Attended Otitis Media: Grade 4 | 0 | 0

22. Secondary Outcome: Serum RSV-neutralizing Antibody Titers and Immunoglobulin G (IgG) Serum Antibody Titers to RSV F Glycoprotein Enzyme-linked Immunosorbent Assay (ELISA) in Subjects (RSV-seronegative) Infected With wt RSV During the RSV Surveillance
Description: Antibodies were assessed by RSV-neutralizing Antibody and Enzyme-linked Immunosorbent Assay (ELISA). A response was defined as a greater than or equal to 4-fold increase in titer in paired specimens, between pre- and post-RSV Surveillance time points.
Time Frame: Measured pre- RSV Surveillance period (baseline) and post-RSV Surveillance period (4-6 months after the baseline)
Population: Only participants who had RSV detected in nasal washes or had greater than or equal to 4 fold rise in serum antibodies from pre- to post-RSV season in the absence of RSV-associated medical events were included.
  Four vaccinees and 3 placebo recipients were excluded due to SARS CoV-2 pandemic and no post-surveillance sample.
Measure: Mean (Standard Deviation); unit: log 2 titers
Arm/Group | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Number analyzed (Participants) | 6 | 4
log 2 titers
  Pre-RSV Surveillance Serum RSV Neutralizing Antibody | 6.7 (1.4) | 3.0 (0.8)
  Post-RSV Surveillance Serum RSV Neutralizing Antibody | 10.7 (1.7) | 8.1 (1.0)
  Pre-RSV Surveillance Serum IgG ELISA RSV F Antibody Interpolated Titers | 10.2 (1.9) | 5.4 (1.7)
  Post-RSV Surveillance Serum IgG ELISA RSV F Antibody Interpolated Titers | 14.3 (1.4) | 11.8 (1.3)

23. Secondary Outcome: Number of Participants With a Greater Than or Equal to 4-fold Rise in Serum RSV-neutralizing Antibody Titers and/or Serum Antibody Titers to RSV F Glycoprotein in RSV-seronegative Subjects (Group 2) Infected With wt RSV During the RSV Surveillance
Description: Serum RSV-neutralizing antibody titers were assessed by 60% RSV-plaque reduction neutralization titer (RSV-PRNT) assay and an Enzyme-linked Immunosorbent Assay (ELISA). Antibody responses were defined as a greater than or equal to 4-fold increase in titer in paired specimens, between pre-RSV surveillance and post-RSV surveillance time points among those who had indicators of natural infection with wt RSV were presented. Natural infection with wt RSV during the RSV season surveillance was defined as having either RSV detected in nasal washes collected during illness visits for MAARI events or a > 4-fold rise in serum antibodies from pre- to post-RSV season in the absence of RSV-associated medical events
Time Frame: Measured pre-RSV Surveillance period (baseline) and post-RSV Surveillance period (4-6 months after the baseline)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
Number analyzed (Participants) | 6 | 4
Participants
  Serum RSV Neutralizing Antibody | 5 | 4
  Serum IgG ELISA RSV F Antibody Interpolated Titers | 6 | 4

ADVERSE EVENTS:
Time Frame: From study entry to end of study. The duration of follow-up for a given participant was 2 months for Group 1 and between 6 and 10 months for Group 2 depending on time of enrollment.
Description: From day 0-28, all SAEs, solicited AEs, and unsolicited AEs, with the exception of the following if not treated with prescription medication or over the counter medications with antipyretic properties: diaper rashes, teething pain, and spitting up. SAEs and LRIs were reported according to Sections 7 & 8 in the Protocol Document. From day 29-56, SAEs were collected. After day 56, from November 1 - March 31 of the following year, medically attended fever, LRI, URI and otitis media were collected.
Arm/Group | Group 1: RSV 6120/∆NS2/1030s Vaccine | Group 1: Placebo | Group 2: RSV 6120/∆NS2/1030s Vaccine | Group 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5 | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5 | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 2/5 | 20/20 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: RSV 6120/∆NS2/1030s Vaccine (N=10) | Group 1: Placebo (N=5) | Group 2: RSV 6120/∆NS2/1030s Vaccine (N=20) | Group 2: Placebo (N=10)
Eye Discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
General Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 9 (16) | 6 (6)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Croup (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 5 (8) | 3 (7)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 9 (14) | 9 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 19 (38) | 8 (16)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT03387137/Prot_SAP_000.pdf
  • Informed Consent Form: RSV-Seronegative (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT03387137/ICF_001.pdf
  • Informed Consent Form: RSV-Seropositive (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT03387137/ICF_002.pdf